CLINICAL TRIAL: NCT00639223
Title: Red Yeast Rice vs. Pravastatin: A Double-Blind Randomized Comparative Study of Myopathic Symptoms
Brief Title: Safety of Red Yeast Rice for High Cholesterol in Individuals With Statin Intolerance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Chestnut Hill Health System (Other)
Responsible Party: David Becker MD Principal Investigator, Chestnut Hill Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 806827
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2009-12

CONDITIONS: Hypercholesterolemia; Statin-Associated Myopathy
Keywords: Statin related myalgia; Hyperlipidemia; Red yeast rice; Cardiovascular Diseases; Nutritional and Metabolic Diseases
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias; Cardiovascular Diseases; Nutritional and Metabolic Diseases | interventions — red yeast rice; Pravastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pravastatin (Active Comparator)
  Interventions: Drug: Pravastatin; Behavioral: Lifestyle modification program
- Red yeast Rice (Experimental)
  Interventions: Dietary Supplement: Red Yeast Rice; Behavioral: Lifestyle modification program

INTERVENTIONS:
Dietary Supplement: Red Yeast Rice — Four 600mg capsules twice daily for 12 weeks
  Arms: Red yeast Rice
Drug: Pravastatin — One 20mg capsule twice daily for 12 weeks
  Other Names: Pravachol
  Arms: Pravastatin
Behavioral: Lifestyle modification program — Weekly sessions each lasting 3 1/2 hours for 12 weeks

SUMMARY:
This study will examine the effect of red yeast rice extract compared to pravastatin on muscle related complaints in individuals with high cholesterol who have previously been unable to tolerate statin medications due to muscle pain. The study will determine whether red yeast is associated with a lower level of muscle related complaints compared to pravastatin.

DETAILED DESCRIPTION:
20 million Americans are actively treated with statins at an annual cost of 16 billion dollars. Statins are effective therapeutic agents for reducing LDL cholesterol and have documented effectiveness. However, a significant subset of patients (5-18%), cannot tolerate lipid lowering statin therapy due to intolerable muscle-related symptoms characterized by muscle pain and/or weakness. These symptoms affect quality of life and lead to poor adherence.

Patients may seek alternative therapies to manage hypercholesterolemia if they have been intolerant of statin therapy. One commonly used alternative treatment option is the Chinese herb red yeast rice extract. Several small studies performed in China, have suggested this treatment is efficacious and well tolerated. In the U.S. red yeast rice is sold over the counter a dietary supplement.

The objective of this study is to critically examine the safety and efficacy of the Chinese herb red yeast rice as an alternative lipid lowering therapy, in a statin intolerant population.

This objective will be operationalized by a double-blind randomized trial, comparing the effect of red yeast rice extract, to that of pravastatin on the level of myalgia in subjects with a prior history of statin-induced myalgias.

The specific aims include:

1. Determine the relative rates of withdrawal from treatment in subjects receiving red yeast rice compared to pravastatin.
2. Determine if red yeast rice is associated with a lower level of muscle pain (myalgia) symptoms compared to pravastatin as measured by the Brief Pain Inventory, a validated pain questionnaire.
3. Determine if red yeast rice is associated with a lower level of muscle weakness compared to pravastatin as measured by a dynamometry, a validated muscle strength testing method.

ELIGIBILITY:
Inclusion Criteria:

* Subject reports stopping at least one statin drug due to complaints of muscle pain or weakness which his/her physician thinks was attributable to the drug.
* Subject has never taken pravastatin.
* Subject willing to remain off the dietary supplements CoQ10, L-carnitine, fish oil, policosanol, and guggulipid, garlic, and phytosterols in margarines (e.g. Benecol, Promise activ), milk or cereal products, for one month prior to the trial and for the duration of the trial.

Exclusion Criteria:

* A history of muscle damage (CK>1000 IU) on statin therapy.
* A history of generalized chronic pain such as fibromyalgia, or generalized arthritis.
* Any active cardiac problem including chest pain, angina, heart attack, bypass surgery, angioplasty/stent or unstable angina/acute coronary syndrome within the past 6 months.
* Taking other lipid lowering drugs including: ezetimibe, gemfibrozil, niacin, fibrates or bile acid sequestrants.
* Triglyceride level more than 400 mg/dl.
* Taking weight loss medication including orlistat, sibutramine, diethylpropion, phendimetrazine, phentermine.
* Taking pain medication or systemic steroids on a chronic basis.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven C Halbert, MD, Study Director — University of Pennsylvania
Locations (1):
- Chestnut Hill Hospital, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pravastatin | Red Yeast Rice
Started | 22 | 21
Completed | 22 | 19
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pravastatin | Red Yeast Rice | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 11 | 25
  >=65 years | 8 | 10 | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 62.9 (6.6) | 62.4 (8.9) | 62.7 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 22 | 21 | 43

OUTCOME MEASURES:

1. Primary Outcome: Withdrawal of Therapy Due to Muscle Symptoms That Are Either Intolerable and/or Associated With a Creatine Kinase(CK) >500
Time Frame: 12 weeks
Measure: Number; unit: Participants
Arm/Group | Pravastatin | Red Yeast Rice
Number analyzed (Participants) | 22 | 21
Participants | 2 | 1

2. Secondary Outcome: Change in LDL-Cholesterol Measured at the Beginning and End of the Study
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Pravastatin | Red Yeast Rice
Number analyzed (Participants) | 22 | 21
Percentage Change | -27.0 (15.4) | -30.2 (10.5)

ADVERSE EVENTS:
Arm/Group | Pravastatin | Red Yeast Rice
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 12/22 | 11/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pravastatin (N=22) | Red Yeast Rice (N=21)
Abdominal bloating or gas (Gastrointestinal disorders) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Small sample size precluded definitive conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No